CLINICAL TRIAL: NCT04818515
Title: A Phase 1b, Open-label, Fixed-sequence, Safety, Tolerability and Drug-drug Interaction Study Between Atogepant and Ubrogepant in Participants With a History of Migraine
Brief Title: Study To Assess Adverse Events and Drug to Drug Interaction of Oral Tablet Atogepant and Ubrogepant in Adult Participants With a History of Migraine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3101-106-002
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Migraine
Keywords: Migraine; Atogepant; Ubrogepant; UBRELVY
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant; ubrogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atogepant, Ubrogepant, and Coadministration (Experimental): Participants will receive oral tablets of ubrogepant, followed be oral tablets of atogepant, followed by administration of oral tablets of atogepant and ubrogepant in combination, for a 30 day interventional period and a 7 day follow up period.
  Interventions: Drug: Atogepant; Drug: Ubrogepant

INTERVENTIONS:
Drug: Atogepant — Oral; Tablet
Drug: Ubrogepant — Oral; Tablet
  Other Names: UBRELVY

SUMMARY:
Migraine is a common neurological disorder typically characterized by attacks of throbbing, moderate to severe headache, often associated with nausea, vomiting, and sensitivity to light and sound. This study will assess the drug to drug interaction between atogepant and ubrogepant and assess the safety of atogepant and ubrogepant, when given alone or in combination, in adult participants with migraine.

Atogepant is an investigational (unapproved) drug for the preventative treatment of migraine. Ubrogepant is a drug approved for the acute treatment of migraine. Adult participants with a history of migraine will be enrolled. Approximately, 30 participants will be enrolled in the study in multiple sites in the United States.

Participants will receive oral tablets of ubrogepant, followed be oral tablets of atogepant, followed by administration of oral tablets of atogepant and ubrogepant in combination. The study duration will be 30 days with a 7 day follow period.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, telephone assessments, blood tests, checking for side effects, and clinician-rated assessments.

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of migraine with or without aura consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd edition (ICHD-3) (2018) and is eligible for preventive migraine treatment.
* By history, the participant's migraines typically last between 4 and 72 hours if untreated or treated unsuccessfully and migraine episodes are separated by at least 48 hours of headache pain freedom.
* History of at least 2 migraine attacks per month in the 2 months prior to screening.
* Sitting heart rate ≥ 45 bpm and ≤ 100 bpm during the vital signs assessment at the Screening Visit. The clinical site may perform a maximum of 2 repeats of vital sign measurements if the initial measurement is out of range.
* Negative test results for benzoylecgonine (cocaine), methadone, barbiturates, amphetamines, benzodiazepines, cannabinoids, opiates, and phencyclidine at the Screening Visit and Day -1; unless explained by concomitant medication use (eg, opioids prescribed for migraine pain).
* Must be a nonsmoker and a nonuser of nicotine-containing products (never smoked or used nicotine-containing products or has not smoked or used nicotine-containing products within the previous 2 years, including eCigarettes).

Exclusion Criteria:

* Difficulty distinguishing migraine headache from tension-type or other headaches.
* Has a history of migraine aura with diplopia or impairment of level of consciousness, hemiplegic migraine, or retinal migraine as defined by ICHD-3.
* Has a current diagnosis of new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or painful cranial neuropathy as defined by ICHD-3.
* Required hospital treatment of a migraine attack 3 or more times in the 6 months prior to screening.
* Has a chronic non-headache pain condition requiring daily pain medication (with the exception of pregabalin).
* Clinically significant cardiovascular or cerebrovascular disease per the investigator's opinion including, but not limited to:

  * Clinically significant ischemic heart disease (eg, unstable angina pectoris).
  * Clinically significant cardiac rhythm or conduction abnormalities (eg, atrial fibrillation, second- or third-degree heart block) or risk factors for torsade de pointes (eg, heart failure, hypokalemia, bradycardia).
  * Myocardial infarction, transient ischemic attack, or stroke within 6 months prior to screening.
  * Heart failure defined as New York Heart Association functional classification system Class III or IV.
* Any clinically significant hematologic, endocrine, pulmonary, renal, hepatic, gastrointestinal, or neurologic disease.
* In the opinion of the investigator, other confounding pain syndromes, confounding psychiatric conditions, dementia, epilepsy, or other significant neurological disorders other than migraine.
* History of malignancy in the 5 years prior to screening, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer.
* History of any prior gastrointestinal conditions (eg, diarrhea syndromes, inflammatory bowel disease) or previous surgery that may affect the absorption or metabolism of study interventions; participants with prior gastric bariatric interventions (eg, Lap Band) which have been reversed are not excluded.
* History of acute hepatitis within 6 months of screening or chronic hepatitis (including nonalcoholic steatohepatitis) or a positive result on anti-human immunodeficiency virus (HIV) type 1 and type 2 antibody, hepatitis B surface antigen (HBsAg), or anti-hepatitis C antibody testing at screening.
* Coronavirus disease 2019 (COVID-19) infection and/or COVID-19 or flu-like symptoms within 14 days of Day 1, including fever, cough, difficulty breathing.
* Close contact with anyone who has a COVID-19 infection within 14 days before Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve from Time 0 to t (AUC0-t), when Ubrogepant is Administered | Day 1
  Area Under the Plasma Concentration-time Curve from 0 to t (AUC0-t), when Ubrogepant is administered.
Area Under the Plasma Concentration-time Curve from Time 0 to t (AUC0-t), when Ubrogepant and Atogepant are Coadministered | Day 1
  Area Under the Plasma Concentration-time Curve from 0 to t (AUC0-t), when ubrogepant and atogepant are coadministered.
Area Under the Plasma Concentration-time Curve from Time 0 to Infinity (AUC0-inf), when Ubrogepant is Administered | Day 1
  Area Under the Plasma Concentration-time Curve from 0 to infinity (AUC0-inf), when Ubrogepant is administered.
Area Under the Plasma Concentration-time Curve from Time 0 to Infinity (AUC0-inf), when when Ubrogepant and Atogepant are Coadministered | Day 1
  Area Under the Plasma Concentration-time Curve from 0 to infinity (AUC0-inf), when ubrogepant and atogepant are coadministered.
Area Under the Plasma Concentration-time Curve During the Dosing Interval at Steady State (AUCtau), when Atogepant is Administered | Day 6
  Area Under the Plasma Concentration-time Curve during the dosing interval at steady state (AUCtau), when Atogepant is administered.
Area Under the Plasma Concentration-time Curve During the Dosing Interval at Steady State (AUCtau), when Ubrogepant and Atogepant are Coadministered | Day 6
  Area Under the Plasma Concentration-time Curve during the dosing interval at steady state (AUCtau), when ubrogepant and atogepant are coadministered.
Maximum Plasma Drug Concentration (Cmax) when Ubrogepant is Administered | Day 1
  Maximum plasma drug concentration (Cmax) when ubrogepant is administered.
Maximum Plasma Drug Concentration (Cmax) when Atogepant is Administered | Day 6
  Maximum plasma drug concentration (Cmax) when atogepant is administered.
Maximum Plasma Drug Concentration (Cmax) of Ubrogepant when Ubrogepant and Atogepant are Coadministered | Day 7
  Maximum plasma drug concentration (Cmax) of ubrogepant when ubrogepant and atogepant are coadministered.
Maximum Plasma Drug Concentration (Cmax) of Atogepant when Ubrogepant and Atogepant are Coadministered | Day 7
  Maximum plasma drug concentration (Cmax) of atogepant when ubrogepant and atogepant are coadministered.

SECONDARY OUTCOMES:
Number of Participants with Abnormal Change in Physical Examinations | Up to Day 28
  Number of participants with abnormal change in physical examinations in areas like cardiovascular, respiratory, gastrointestinal, and neurological systems will be assessed.
Number of Participants with Abnormal Change From Baseline in Vital Sign Measurements | Up to Day 28
  Number of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Number of Participants with Abnormal Change in Clinical Laboratory Test Results Like Hematology will be Assessed | Up to Day 28
  Number of participants with abnormal change in clinical laboratory test results like hematology will be assessed.
Change From Baseline in Electrocardiograms (ECGs) | Up to Day 28
  12-lead resting ECGs will be recorded. Parameters include heart rate, PR interval, QT interval, QRS duration, and QT interval corrected using Fridericia's formula (QTcF).
Change from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Day 29
  The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior, with a higher score denoting more severe suicidal ideation and behavior.
Number of Participants with Adverse Events (AE) | Up to Day 37
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (3):
  - PPD Clinical Research Unit /ID# 227676, Orlando, Florida
  - Bio-Kinetic Clinical Applications, LLC /ID# 227675, Springfield, Missouri
  - Spaulding Clinical Research LLC /ID# 229505, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=3101-106-002&Latitude=&Longitude=&LocationName=#additional-resources-section